CLINICAL TRIAL: NCT00483613
Title: Effects of Treatment of Chronic Stress in Patients With Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Virgen de las Nieves (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-Alonso
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2007-06-07 (Estimated); Status verified 2007-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Daily stress; Cognitive-behavioral therapy; Quality of life; SLEDAI
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy of Meichenbaum

SUMMARY:
* Daily stress can worsens the clinical course of lupus.
* Objective: to determine the efficacy of the stress management therapy in a group of patients with lupus.
* 45 patients with lupus and high daily stress participated in this clinical trial.
* Two groups resulted: a control group (CG) that received the usual care and a therapy group (TG) that received a cognitive behavioral therapy.
* The therapy consisted of ten consecutive weekly sessions.
* The measured variables were psychological, clinical, immunological and quality of life. At the basal moment and after 3, 9 and 15 months.
* Statistical analysis showed a significant reduction in the levels of depression, anxiety and daily stress in the therapy group, compared to the usual care group, a significant improvement in quality of life, improvements in the reported symptoms (cardiovascular, respiratory, cutaneous and musculoskeletal.

DETAILED DESCRIPTION:
Stress, especially daily stress, worsens the lupus symptoms perceived by the patients. Our objective was to determine the efficacy of the Meichenbaum stress management therapy for dealing with high daily stress in a group of patients with lupus.

We designed a randomized clinical trial in which 45 patients with lupus and daily stress participated. The patients were randomly assigned to one of the following groups: a) a control group (CG) that received the usual care and b) a therapy group (TG) that received a cognitive behavioral type therapy, performed by a group of 3 psychologists. Both groups were similar with regard to their sociodemographic, clinical, immunological, psychological aspects at the basal moment. The therapy consisted of ten consecutive weekly sessions. Psychological and emotional, clinical, immunological variables and quality of life were evaluated at the basal moment and after 3, 9 and 15 months.

The between-groups analysis showed a significant reduction in the levels of depression, anxiety and daily stress in the TG, compared to the CG, throughout the entire follow-up period, as well as a significant improvement in quality of life. The results also showed improvements in the reported symptoms (cardiovascular, respiratory, cutaneous and musculoskeletal) in the patients from the TG, who showed significant differences with regard to their basal level and in comparison with CG patients. This study shows the efficacy of the Meichenbaum stress management therapy in patients with lupus and high daily stress, as it significantly reduces the incidence of psychological disorders related to suffering from lupus, and it significantly improves and maintains their quality of life, in spite of the absence of a significant reduction in the illness activity index.

ELIGIBILITY:
Inclusion Criteria:

* SLE with at least 4 ACR criteria or patients with a diagnosis of CCL made with a biopsy
* over 18 years of age
* high levels of daily stress (defined in our population as equal to or greater than 24 points for men and 27 for women on the Cohen Perceived Stress Scale)

Exclusion Criteria:

* less than a year of diagnosis of the disease
* illiteracy
* not being available to attend the intervention sessions or to perform the established analytic determinations
* treatment for an acute psychiatric pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-12; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Activity of the disease, quality of life | Initial, 3rd. month, 9th month, 15 th month

SECONDARY OUTCOMES:
Vulnerability to stress, amount of stress, depression, anxiety, SLEDAI index activity of lupus, somatic symptoms, number of clinical flares, antiADNn antibodies and levels of seric complement C3 and C4 | Initial, 3rd month, 9th month, 15th month

CONTACTS AND LOCATIONS:
Overall Officials: Jiménez Juan, PhD, MD, Principal Investigator
Locations (1):
- University Hospital Virgen de las Nieves, Granada, Spain/Granada, Spain

REFERENCES:
- [Background] Peralta-Ramirez MI, Jimenez-Alonso J, Godoy-Garcia JF, Perez-Garcia M; Group Lupus Virgen de las Nieves. The effects of daily stress and stressful life events on the clinical symptomatology of patients with lupus erythematosus. Psychosom Med. 2004 Sep-Oct;66(5):788-94. doi: 10.1097/01.psy.0000133327.41044.94. PMID 15385708
- [Result] Peralta-Ramirez MI, Coin-Mejias MA, Jimenez-Alonso J, Ortego-Centeno N, Callejas-Rubio JL, Caracuel-Romero A, Perez-Garcia M. Stress as a predictor of cognitive functioning in lupus. Lupus. 2006;15(12):858-64. doi: 10.1177/0961203306071404. PMID 17211991